CLINICAL TRIAL: NCT07169123
Title: Protease Regulation and Impact of Sodium as Mechanisms of Inflammation in IBD
Acronym: PRISM-IBD
Status: Not yet recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, David Armstrong, Principal Investigator, McMaster University
Other Study IDs: HiREB-18816
Record Dates: First submitted 2025-06-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Crohns Disease
Keywords: sodium; Crohn's disease; proteases; diet
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The following samples will be retained for analysis: blood (for sodium, CRP, and metabolomics), stool (for microbiota, metabolomics, fecal calprotectin, and proteolytic activity), and spot urine (for sodium, creatinine, potassium, and metabolomics). In Phase 2, additional fecal samples will be collected for microbiota and metabolomics analysis, along with blood and urine (for metabolomics), and colonic biopsies (for microbiota composition, metabolomics, proteolytic activity, and microbial proteases).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study looks at how eating salt affects gut health in people with Crohn's disease. The aim of the study is to find out whether eating more salt increases the breakdown of proteins in the gut and if this makes inflammation and symptoms worse. By studying the link between salt, gut bacteria and inflammation, the study hopes to improve diet advice for people with Crohn's disease. This research may help find specific foods that affect the disease and lead to better, more personalized nutrition plans.

DETAILED DESCRIPTION:
This longitudinal exploratory study has two related phases:

Phase 1 will enroll 300 Crohn's disease (CD) patients from McMaster's IBD and IBD Nutrition Clinics to assess dietary sodium intake and fecal proteolytic activity in relation to disease activity (active/inactive). Participants will be followed annually for 2 years, forming a registry. At baseline and each follow-up visit, data collected will include: demographics, BMI, CDAI, diet (1-week food recall via Keenoa and 6-month sodium questionnaire), blood (sodium, metabolomics, CRP), stool (microbiota, metabolomics, fecal calprotectin, proteolytic activity), and spot urine (sodium, potassium, creatinine, metabolomics). Extra visits will occur if a disease flare happens.

Phase 2 will involve 80 participants from Phase 1 (40 high-sodium diet [HSD], 40 low-sodium diet [LSD]), selected based on sodium intake. Over three visits (baseline, week 1, week 2), participants will provide fecal samples for microbiota and metabolomics analysis, and blood/urine samples (baseline and week 2). Colonoscopy with biopsies and video will be performed at week 2. Diet will be closely tracked using Keenoa to assess intake of sodium, carbs, UPF, fibre, and calories. After Phase 2, participants return to Phase 1 follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 70 years of age
* Crohn's disease diagnosis
* Willing and able to sign written informed consent prior to study entry
* Able to comply with the study procedures, in the opinion of the investigator

Exclusion Criteria:

* Antibiotics, antibacterial agents, or probiotics, currently, or within the last 8 weeks
* Alcohol or drug abuse
* Pregnancy
* Concurrent systemic disease and/or laboratory abnormalities considered by investigators to be a risk or that could interfere with data collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Crohn's disease followed at McMaster University's Gastroenterology Outpatient Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Dietary Sodium Intake | Phase 1: baseline (Year 0); Year 1; and Year 2. Phase 2: baseline (Week 0); Week 1; and Week 2.
  Dietary sodium intake will be assessed via 24-hour dietary recall and sodium-specific food frequency questionnaires (mg/day). Values will be used to classify participants as HSD or LSD and correlated with changes in proteolytic activity, mucosal permeability, and disease activity.

SECONDARY OUTCOMES:
Proteolytic Activity in Stool and Colonic Biopsies | Stool: Phase 1 - baseline (Year 0); Year 1; and Year 2. Biopsy: Phase 2 - Week 2
  Proteolytic activity will be assessed in fecal samples and colonic biopsies. Fecal samples will be analyzed for host and bacterial proteases (units of proteolytic activity per gram of stool, U/g), and colonic biopsies for host and bacterial proteases (units of proteolytic activity per mg of tissue, U/mg). Comparisons will be made between participants consuming a high-sodium diet (HSD) and a low-sodium diet (LSD) to evaluate associations with mucosal barrier dysfunction and disease activity over time.
Crohn's Disease Activity Index (CDAI) | Phase 1: baseline (Year 0); Year 1; and Year 2. Phase 2: baseline (Week 0); and Week 2.
  Crohn's Disease Activity Index will be calculated using patient-reported symptoms, physical exam findings, and lab values (score, unitless). CDAI <150 indicates remission, 150-220 mild disease, 220-450 moderate disease, and >450 severe disease. CDAI scores will be compared between HSD and LSD groups to evaluate changes in clinical disease activity over time.
Mucosal Permeability | Phase 2: Week 2
  Colonic biopsies will be analyzed for mucosal barrier integrity using permeability assays (e.g., FITC-dextran flux). Higher values indicate greater barrier dysfunction (permeability index, arbitrary units). Comparisons will be made between HSD and LSD groups to determine effects of dietary sodium intake.
Patient Subgroup Characterization Based on Metabolic and Microbial Profiles | Phase 1: baseline (Year 0); Year 1; and Year 2. Phase 2: baseline (Week 0); Week 1; and Week 2.
  Participants will be characterized using dietary sodium intake, metabolic profiling (blood, urine, stool), and microbial activity (stool and biopsy-based proteolytic and microbiome analyses). Data will identify subgroups with distinct metabolic signatures, sodium intake levels, microbial profiles, and disease progression, providing insight into diet-microbiota-host metabolism interactions in Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Pang Z, Lu Y, Zhou G, Hui F, Xu L, Viau C, Spigelman AF, MacDonald PE, Wishart DS, Li S, Xia J. MetaboAnalyst 6.0: towards a unified platform for metabolomics data processing, analysis and interpretation. Nucleic Acids Res. 2024 Jul 5;52(W1):W398-W406. doi: 10.1093/nar/gkae253. PMID 38587201
- [Background] Caminero A, Herran AR, Nistal E, Perez-Andres J, Vaquero L, Vivas S, Ruiz de Morales JM, Albillos SM, Casqueiro J. Diversity of the cultivable human gut microbiome involved in gluten metabolism: isolation of microorganisms with potential interest for coeliac disease. FEMS Microbiol Ecol. 2014 May;88(2):309-19. doi: 10.1111/1574-6941.12295. Epub 2014 Mar 3. PMID 24499426
- [Background] Whelan FJ, Waddell B, Syed SA, Shekarriz S, Rabin HR, Parkins MD, Surette MG. Culture-enriched metagenomic sequencing enables in-depth profiling of the cystic fibrosis lung microbiota. Nat Microbiol. 2020 Feb;5(2):379-390. doi: 10.1038/s41564-019-0643-y. Epub 2020 Jan 20. PMID 31959969
- [Background] Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. Genome Biol. 2014;15(12):550. doi: 10.1186/s13059-014-0550-8. PMID 25516281
- [Background] Paulson JN, Stine OC, Bravo HC, Pop M. Differential abundance analysis for microbial marker-gene surveys. Nat Methods. 2013 Dec;10(12):1200-2. doi: 10.1038/nmeth.2658. Epub 2013 Sep 29. PMID 24076764
- [Background] Buchfink B, Xie C, Huson DH. Fast and sensitive protein alignment using DIAMOND. Nat Methods. 2015 Jan;12(1):59-60. doi: 10.1038/nmeth.3176. Epub 2014 Nov 17. PMID 25402007
- [Background] Bushnell B, Rood J, Singer E. BBMerge - Accurate paired shotgun read merging via overlap. PLoS One. 2017 Oct 26;12(10):e0185056. doi: 10.1371/journal.pone.0185056. eCollection 2017. PMID 29073143
- [Background] Kopylova E, Noe L, Touzet H. SortMeRNA: fast and accurate filtering of ribosomal RNAs in metatranscriptomic data. Bioinformatics. 2012 Dec 15;28(24):3211-7. doi: 10.1093/bioinformatics/bts611. Epub 2012 Oct 15. PMID 23071270
- [Background] Kim D, Paggi JM, Park C, Bennett C, Salzberg SL. Graph-based genome alignment and genotyping with HISAT2 and HISAT-genotype. Nat Biotechnol. 2019 Aug;37(8):907-915. doi: 10.1038/s41587-019-0201-4. Epub 2019 Aug 2. PMID 31375807
- [Background] Kang DD, Li F, Kirton E, Thomas A, Egan R, An H, Wang Z. MetaBAT 2: an adaptive binning algorithm for robust and efficient genome reconstruction from metagenome assemblies. PeerJ. 2019 Jul 26;7:e7359. doi: 10.7717/peerj.7359. eCollection 2019. PMID 31388474
- [Background] Nurk S, Meleshko D, Korobeynikov A, Pevzner PA. metaSPAdes: a new versatile metagenomic assembler. Genome Res. 2017 May;27(5):824-834. doi: 10.1101/gr.213959.116. Epub 2017 Mar 15. PMID 28298430
- [Background] Moayyedi P, MacQueen G, Bernstein CN, Vanner S, Bercik P, Madsen KL, Surette M, Rioux JD, Dieleman LA, Verdu E, de Souza RJ, Otley A, Targownik L, Lavis J, Cunningham J, Marshall DA, Zelinsky S, Fernandes A. IMAGINE Network's Mind And Gut Interactions Cohort (MAGIC) Study: a protocol for a prospective observational multicentre cohort study in inflammatory bowel disease and irritable bowel syndrome. BMJ Open. 2020 Oct 21;10(10):e041733. doi: 10.1136/bmjopen-2020-041733. PMID 33087380
- [Background] Franzosa EA, McIver LJ, Rahnavard G, Thompson LR, Schirmer M, Weingart G, Lipson KS, Knight R, Caporaso JG, Segata N, Huttenhower C. Species-level functional profiling of metagenomes and metatranscriptomes. Nat Methods. 2018 Nov;15(11):962-968. doi: 10.1038/s41592-018-0176-y. Epub 2018 Oct 30. PMID 30377376
- [Background] Segata N, Waldron L, Ballarini A, Narasimhan V, Jousson O, Huttenhower C. Metagenomic microbial community profiling using unique clade-specific marker genes. Nat Methods. 2012 Jun 10;9(8):811-4. doi: 10.1038/nmeth.2066. PMID 22688413
- [Background] Langmead B, Salzberg SL. Fast gapped-read alignment with Bowtie 2. Nat Methods. 2012 Mar 4;9(4):357-9. doi: 10.1038/nmeth.1923. PMID 22388286
- [Background] Chen S, Zhou Y, Chen Y, Gu J. fastp: an ultra-fast all-in-one FASTQ preprocessor. Bioinformatics. 2018 Sep 1;34(17):i884-i890. doi: 10.1093/bioinformatics/bty560. PMID 30423086
- [Background] Derakhshani H, Bernier SP, Marko VA, Surette MG. Completion of draft bacterial genomes by long-read sequencing of synthetic genomic pools. BMC Genomics. 2020 Jul 29;21(1):519. doi: 10.1186/s12864-020-06910-6. PMID 32727443
- [Background] Kanehisa M, Goto S. KEGG: kyoto encyclopedia of genes and genomes. Nucleic Acids Res. 2000 Jan 1;28(1):27-30. doi: 10.1093/nar/28.1.27. PMID 10592173
- [Background] Douglas GM, Maffei VJ, Zaneveld JR, Yurgel SN, Brown JR, Taylor CM, Huttenhower C, Langille MGI. PICRUSt2 for prediction of metagenome functions. Nat Biotechnol. 2020 Jun;38(6):685-688. doi: 10.1038/s41587-020-0548-6. No abstract available. PMID 32483366
- [Background] Langille MG, Zaneveld J, Caporaso JG, McDonald D, Knights D, Reyes JA, Clemente JC, Burkepile DE, Vega Thurber RL, Knight R, Beiko RG, Huttenhower C. Predictive functional profiling of microbial communities using 16S rRNA marker gene sequences. Nat Biotechnol. 2013 Sep;31(9):814-21. doi: 10.1038/nbt.2676. Epub 2013 Aug 25. PMID 23975157
- [Background] McMurdie PJ, Holmes S. phyloseq: an R package for reproducible interactive analysis and graphics of microbiome census data. PLoS One. 2013 Apr 22;8(4):e61217. doi: 10.1371/journal.pone.0061217. Print 2013. PMID 23630581
- [Background] Price MN, Dehal PS, Arkin AP. FastTree 2--approximately maximum-likelihood trees for large alignments. PLoS One. 2010 Mar 10;5(3):e9490. doi: 10.1371/journal.pone.0009490. PMID 20224823
- [Background] Quast C, Pruesse E, Yilmaz P, Gerken J, Schweer T, Yarza P, Peplies J, Glockner FO. The SILVA ribosomal RNA gene database project: improved data processing and web-based tools. Nucleic Acids Res. 2013 Jan;41(Database issue):D590-6. doi: 10.1093/nar/gks1219. Epub 2012 Nov 28. PMID 23193283
- [Background] Callahan BJ, McMurdie PJ, Rosen MJ, Han AW, Johnson AJ, Holmes SP. DADA2: High-resolution sample inference from Illumina amplicon data. Nat Methods. 2016 Jul;13(7):581-3. doi: 10.1038/nmeth.3869. Epub 2016 May 23. PMID 27214047
- [Background] Bolger AM, Lohse M, Usadel B. Trimmomatic: a flexible trimmer for Illumina sequence data. Bioinformatics. 2014 Aug 1;30(15):2114-20. doi: 10.1093/bioinformatics/btu170. Epub 2014 Apr 1. PMID 24695404
- [Background] Constante M, Libertucci J, Galipeau HJ, Szamosi JC, Rueda G, Miranda PM, Pinto-Sanchez MI, Southward CM, Rossi L, Fontes ME, Chirdo FG, Surette MG, Bercik P, Caminero A, Verdu EF. Biogeographic Variation and Functional Pathways of the Gut Microbiota in Celiac Disease. Gastroenterology. 2022 Nov;163(5):1351-1363.e15. doi: 10.1053/j.gastro.2022.06.088. Epub 2022 Jul 8. PMID 35810781
- [Background] Szamosi JC, Forbes JD, Copeland JK, Knox NC, Shekarriz S, Rossi L, Graham M, Bonner C, Guttman DS, Van Domselaar G, Surette MG, Bernstein CN. Assessment of Inter-Laboratory Variation in the Characterization and Analysis of the Mucosal Microbiota in Crohn's Disease and Ulcerative Colitis. Front Microbiol. 2020 Aug 21;11:2028. doi: 10.3389/fmicb.2020.02028. eCollection 2020. PMID 32973734
- [Background] Mason B, Ross L, Gill E, Healy H, Juffs P, Kark A. Development and validation of a dietary screening tool for high sodium consumption in Australian renal patients. J Ren Nutr. 2014 Mar;24(2):123-34.e1-3. doi: 10.1053/j.jrn.2013.10.004. Epub 2014 Jan 3. PMID 24394445
- [Background] Ji Y, Plourde H, Bouzo V, Kilgour RD, Cohen TR. Validity and Usability of a Smartphone Image-Based Dietary Assessment App Compared to 3-Day Food Diaries in Assessing Dietary Intake Among Canadian Adults: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Sep 9;8(9):e16953. doi: 10.2196/16953. PMID 32902389
- [Background] Brown IJ, Dyer AR, Chan Q, Cogswell ME, Ueshima H, Stamler J, Elliott P; INTERSALT Co-Operative Research Group. Estimating 24-hour urinary sodium excretion from casual urinary sodium concentrations in Western populations: the INTERSALT study. Am J Epidemiol. 2013 Jun 1;177(11):1180-92. doi: 10.1093/aje/kwt066. Epub 2013 May 14. PMID 23673246
- [Background] Lahiff C, Safaie P, Awais A, Akbari M, Gashin L, Sheth S, Lembo A, Leffler D, Moss AC, Cheifetz AS. The Crohn's disease activity index (CDAI) is similarly elevated in patients with Crohn's disease and in patients with irritable bowel syndrome. Aliment Pharmacol Ther. 2013 Apr;37(8):786-94. doi: 10.1111/apt.12262. Epub 2013 Feb 21. PMID 23432394
- [Background] Gracie DJ, Williams CJ, Sood R, Mumtaz S, Bholah MH, Hamlin PJ, Ford AC. Poor Correlation Between Clinical Disease Activity and Mucosal Inflammation, and the Role of Psychological Comorbidity, in Inflammatory Bowel Disease. Am J Gastroenterol. 2016 Apr;111(4):541-51. doi: 10.1038/ajg.2016.59. Epub 2016 Mar 22. PMID 27002800
- [Background] Jukic A, Bakiri L, Wagner EF, Tilg H, Adolph TE. Calprotectin: from biomarker to biological function. Gut. 2021 Oct;70(10):1978-1988. doi: 10.1136/gutjnl-2021-324855. Epub 2021 Jun 18. PMID 34145045
- [Background] Arcand J, Floras JS, Azevedo E, Mak S, Newton GE, Allard JP. Evaluation of 2 methods for sodium intake assessment in cardiac patients with and without heart failure: the confounding effect of loop diuretics. Am J Clin Nutr. 2011 Mar;93(3):535-41. doi: 10.3945/ajcn.110.004457. Epub 2010 Dec 29. PMID 21191141
- [Background] Miranda PM, De Palma G, Serkis V, Lu J, Louis-Auguste MP, McCarville JL, Verdu EF, Collins SM, Bercik P. High salt diet exacerbates colitis in mice by decreasing Lactobacillus levels and butyrate production. Microbiome. 2018 Mar 22;6(1):57. doi: 10.1186/s40168-018-0433-4. PMID 29566748
- [Background] Vergnolle N. Protease inhibition as new therapeutic strategy for GI diseases. Gut. 2016 Jul;65(7):1215-24. doi: 10.1136/gutjnl-2015-309147. Epub 2016 Apr 12. PMID 27196587
- [Background] Galipeau HJ, Caminero A, Turpin W, Bermudez-Brito M, Santiago A, Libertucci J, Constante M, Raygoza Garay JA, Rueda G, Armstrong S, Clarizio A, Smith MI, Surette MG, Bercik P; CCC Genetics, Environmental, Microbial Project Research Consortium; Croitoru K, Verdu EF. Novel Fecal Biomarkers That Precede Clinical Diagnosis of Ulcerative Colitis. Gastroenterology. 2021 Apr;160(5):1532-1545. doi: 10.1053/j.gastro.2020.12.004. Epub 2020 Dec 10. PMID 33310084
- [Background] Pittayanon R, Lau JT, Leontiadis GI, Tse F, Yuan Y, Surette M, Moayyedi P. Differences in Gut Microbiota in Patients With vs Without Inflammatory Bowel Diseases: A Systematic Review. Gastroenterology. 2020 Mar;158(4):930-946.e1. doi: 10.1053/j.gastro.2019.11.294. Epub 2019 Dec 5. PMID 31812509
- [Background] Lopez-Siles M, Enrich-Capo N, Aldeguer X, Sabat-Mir M, Duncan SH, Garcia-Gil LJ, Martinez-Medina M. Alterations in the Abundance and Co-occurrence of Akkermansia muciniphila and Faecalibacterium prausnitzii in the Colonic Mucosa of Inflammatory Bowel Disease Subjects. Front Cell Infect Microbiol. 2018 Sep 7;8:281. doi: 10.3389/fcimb.2018.00281. eCollection 2018. PMID 30245977
- [Background] Machiels K, Joossens M, Sabino J, De Preter V, Arijs I, Eeckhaut V, Ballet V, Claes K, Van Immerseel F, Verbeke K, Ferrante M, Verhaegen J, Rutgeerts P, Vermeire S. A decrease of the butyrate-producing species Roseburia hominis and Faecalibacterium prausnitzii defines dysbiosis in patients with ulcerative colitis. Gut. 2014 Aug;63(8):1275-83. doi: 10.1136/gutjnl-2013-304833. Epub 2013 Sep 10. PMID 24021287
- [Background] Lo CH, Khandpur N, Rossato SL, Lochhead P, Lopes EW, Burke KE, Richter JM, Song M, Ardisson Korat AV, Sun Q, Fung TT, Khalili H, Chan AT, Ananthakrishnan AN. Ultra-processed Foods and Risk of Crohn's Disease and Ulcerative Colitis: A Prospective Cohort Study. Clin Gastroenterol Hepatol. 2022 Jun;20(6):e1323-e1337. doi: 10.1016/j.cgh.2021.08.031. Epub 2021 Aug 28. PMID 34461300
- [Background] Chen J, Wellens J, Kalla R, Fu T, Deng M, Zhang H, Yuan S, Wang X, Theodoratou E, Li X, Satsangi J. Intake of Ultra-processed Foods Is Associated with an Increased Risk of Crohn's Disease: A Cross-sectional and Prospective Analysis of 187 154 Participants in the UK Biobank. J Crohns Colitis. 2023 Apr 19;17(4):535-552. doi: 10.1093/ecco-jcc/jjac167. PMID 36305857
- [Background] Vagianos K, Dolovich C, Witges K, Graff LA, Bernstein CN. Ultra-Processed Food, Disease Activity, and Inflammation in Ulcerative Colitis: The Manitoba Living With IBD Study. Am J Gastroenterol. 2024 Jun 1;119(6):1102-1109. doi: 10.14309/ajg.0000000000002667. Epub 2024 Feb 2. PMID 38305329
- [Background] Narula N, Wong ECL, Dehghan M, Mente A, Rangarajan S, Lanas F, Lopez-Jaramillo P, Rohatgi P, Lakshmi PVM, Varma RP, Orlandini A, Avezum A, Wielgosz A, Poirier P, Almadi MA, Altuntas Y, Ng KK, Chifamba J, Yeates K, Puoane T, Khatib R, Yusuf R, Bostrom KB, Zatonska K, Iqbal R, Weida L, Yibing Z, Sidong L, Dans A, Yusufali A, Mohammadifard N, Marshall JK, Moayyedi P, Reinisch W, Yusuf S. Association of ultra-processed food intake with risk of inflammatory bowel disease: prospective cohort study. BMJ. 2021 Jul 14;374:n1554. doi: 10.1136/bmj.n1554. PMID 34261638
- [Background] Christ A, Lauterbach M, Latz E. Western Diet and the Immune System: An Inflammatory Connection. Immunity. 2019 Nov 19;51(5):794-811. doi: 10.1016/j.immuni.2019.09.020. PMID 31747581
- [Background] Windsor JW, Kuenzig ME, Murthy SK, Bitton A, Bernstein CN, Jones JL, Lee K, Targownik LE, Pena-Sanchez JN, Rohatinsky N, Ghandeharian S, Im JHB, Davis T, Weinstein J, Goddard Q, Benchimol EI, Kaplan GG. The 2023 Impact of Inflammatory Bowel Disease in Canada: Executive Summary. J Can Assoc Gastroenterol. 2023 Jun 1;6(Suppl 2):S1-S8. doi: 10.1093/jcag/gwad003. eCollection 2023 Sep. PMID 37674500
- [Background] Gisbert JP, Chaparro M. Primary Failure to an Anti-TNF Agent in Inflammatory Bowel Disease: Switch (to a Second Anti-TNF Agent) or Swap (for Another Mechanism of Action)? J Clin Med. 2021 Nov 15;10(22):5318. doi: 10.3390/jcm10225318. PMID 34830595